CLINICAL TRIAL: NCT02776267
Title: Percutaneous Coronary Intervention With the ANgiolite Drug-Eluting Stent: an Optical CoHerence TOmogRaphy Study. The ANCHOR Study
Brief Title: Percutaneous Coronary Intervention With the Angiolite Drug-eluting Stent: an Optical Cohenrece Tomography Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josep Rodes-Cabau (Other)
Collaborators: iVascular (Unknown)
Responsible Party: Sponsor-Investigator, Josep Rodes-Cabau, MD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANCHOR
Record Dates: First submitted 2016-02-07; First posted 2016-05-18 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Angiolite stent - 3-month angiogram/OCT (Experimental): Patients scheduled for PCI (and whot meet pre-specified inlcusion criteria) are enrolled to receive the Angiolite DES. They will undergo a scheduled repeat coronary angiogram and OCT evaluation at 3-month post index PCI.
  Interventions: Device: Angiolite stent
- Angiolite stent - 6-month angiogram/OCT (Experimental): Patients scheduled for PCI (and whot meet pre-specified inlcusion criteria) are enrolled to receive the Angiolite DES. They will undergo a scheduled repeat coronary angiogram and OCT evaluation at 6-month post index PCI.
  Interventions: Device: Angiolite stent

INTERVENTIONS:
Device: Angiolite stent — Following index PCI, patients will be followed via scheduled clinic and/or phone contact at 1-, 3-, 6-, 12- and 24-month. Patient will be randomized to undergo a scheduled repeat coronary angiogram and OCT evaluation at either at 3- or 6-month post index PCI.
  Other Names: (Angiolite CE Mark reference number: 2014 12 0833 ED)

SUMMARY:
The purpose of this study is to perform a first-in-man assessment of feasibility, exploratory efficacy and clinical performance of the novel Angiolite drug-eluting stent (iVascular, Barcelona, Spain) utilizing intracoronary optical coherence tomography (OCT).

DETAILED DESCRIPTION:
This is a prospective registry including patient scheduled for a clinically-indicated percutaneous coronary intervention (PCI) of a de novo epicardial lesion with indication for drug-eluting stent implantation. Following study enrolment and PCI/stent with the Angiolite DES, patients will be scheduled for follow-up surveillance coronary angiography and OCT with the C7-XRTM Fourier Domain OCT system with C7 DragonflyTM catheter (St Jude Medical, Minneapolis, MN) or with the Terumo LunawayTM OCT system with fastview catheter (Terumo Medical Corporation, Tokyo, Japan). An adaptive design component of the study will randomize patients to either 3-month or 6-month angio/OCT follow-up. Clinical follow-up will occur at 30 days, 3 months, 6 months, 12 months and 24 months post PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for clinically-indicated PCI of a de nove epicardial lesion, including those with chronic stable angina, ACS (defined as NSTEMI or ACS with negative cardiac enzymes) or in the setting of elective PCI.
* Indication for DES implantation
* Target lesion must have visually estimated stenosis ≥50% and one of the following: stenosis ≥70% or evidence of ischemia
* Strong preference for single stent coverage per lesion, but if unexpected clinically indicated second stent placement with overlap is needed, these patients will not be excluded from optical coherence tomographic follow-up
* Target lesion, if possible, should be predilated/pretreated

Exclusion Criteria:

* Age >85 years
* Acute ST segment elevation MI (STEMI)
* Cardiogenic shock
* Known left ventricular ejection fraction <30%
* Contraindication for dual antiplatelet therapy (DAPT) for at least 6-month duration
* Iodinated contrast allergy
* Renal impairment with serum creatinine >2.0 mg/dL
* Anticipated medical non-compliance
* Life-expectancy <12 months
* Chronic total occlusion (CTO) in the target vessel
* Bifurcation lesion requiring a two-stent strategy
* In-stent restenosis
* Severe lesion/segment angulation/tortuosity
* Severe vessel/lesion calcification
* Simultaneous PCI within the same or different vessel during the same procedure
* Lesion unsuitable for OCT (proximal lesions <10 mm from ostium of left main or right coronary arteries)
* Lesion length >18 mm
* Stent length >24 mm
* Stent diameter ≤2.5 mm and > 4.0 mm
* Unprotected left main coronary artery disease (≥50% diameter stenosis)
* >1 lesion
* Planned use of 2 overlapping stents

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Neo-intimal coverage | 6-month
  Strut-based analysis: % of covered struts. Cross-sectional analysis: number of cross-sections with RUTTS (Rate of uncovered to total number of struts) score>30%.
  Measured by an independant OCT laboratory
Neo-intimal obstruction | 6-month
  Strut-based analysis: mean neointimal thickness (µm). Cross-sectional analysis: neointimal volume obstruction (%). Measured by an independant OCT laboratory

SECONDARY OUTCOMES:
Neo-intimal coverage | 3-month
  Strut-based analysis: % of covered struts. Cross-sectional analysis: number of cross-sections with RUTTS (Rate of uncovered to total number of struts) score>30%.
  Measured by an independant OCT laboratory.
Neo-intimal obstruction | 3-month
  Strut-based analysis: mean neointimal thickness (µm). Cross-sectional analysis: neointimal volume obstruction (%). Measured by an independant OCT laboratory.
Apposition | 3- and 6-month
  Strut-based analysis: incomplete strut apposition (ISA) rate. Cross-sectional analysis: % frames with ISA. Measured by an independant OCT laboratory.
In-stent angiographic late lumen in mm | 6-month
  Confirmed by Imaging and measured by an independant QCA laboratory
In-stent and in-segment restenosis | 6-month
  Confirmed by Imaging and measured by an independant QCA laboratory (Reduction in percent diameter stenosis of stented segment of >= 50%
CV death | 6-month and 1-year
  Death from any known cardiovascular etiology
Myocardial infarction | Peri-procedural, spontaneous
  Peri-procedural myocardial infarction will be defined according to the 3rd universal definition of MI Following PCI, myocardial infarction will be defined according to the specific clinical situation of the patient.
Target-lesion revascularization | 24 months
  Any repeat revascularization du to a restenosis within the DES-treated segment
Binary restenosis | 24 months
  Reduction in percent diameter stenosis of stented segment of < vs.>= 50%

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodes-Cabau, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (4):
- Spain (4):
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Universitario de Leon, León
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farooq V, Gogas BD, Serruys PW. Restenosis: delineating the numerous causes of drug-eluting stent restenosis. Circ Cardiovasc Interv. 2011 Apr 1;4(2):195-205. doi: 10.1161/CIRCINTERVENTIONS.110.959882. No abstract available. PMID 21505166
- [Background] Garg S, Serruys PW. Coronary stents: current status. J Am Coll Cardiol. 2010 Aug 31;56(10 Suppl):S1-42. doi: 10.1016/j.jacc.2010.06.007. PMID 20797502
- [Background] Daemen J, Wenaweser P, Tsuchida K, Abrecht L, Vaina S, Morger C, Kukreja N, Juni P, Sianos G, Hellige G, van Domburg RT, Hess OM, Boersma E, Meier B, Windecker S, Serruys PW. Early and late coronary stent thrombosis of sirolimus-eluting and paclitaxel-eluting stents in routine clinical practice: data from a large two-institutional cohort study. Lancet. 2007 Feb 24;369(9562):667-78. doi: 10.1016/S0140-6736(07)60314-6. PMID 17321312
- [Background] Nakazawa G, Finn AV, Joner M, Ladich E, Kutys R, Mont EK, Gold HK, Burke AP, Kolodgie FD, Virmani R. Delayed arterial healing and increased late stent thrombosis at culprit sites after drug-eluting stent placement for acute myocardial infarction patients: an autopsy study. Circulation. 2008 Sep 9;118(11):1138-45. doi: 10.1161/CIRCULATIONAHA.107.762047. Epub 2008 Aug 25. PMID 18725485
- [Background] Serruys PW, Ormiston JA, Onuma Y, Regar E, Gonzalo N, Garcia-Garcia HM, Nieman K, Bruining N, Dorange C, Miquel-Hebert K, Veldhof S, Webster M, Thuesen L, Dudek D. A bioabsorbable everolimus-eluting coronary stent system (ABSORB): 2-year outcomes and results from multiple imaging methods. Lancet. 2009 Mar 14;373(9667):897-910. doi: 10.1016/S0140-6736(09)60325-1. PMID 19286089
- [Background] Prati F, Guagliumi G, Mintz GS, Costa M, Regar E, Akasaka T, Barlis P, Tearney GJ, Jang IK, Arbustini E, Bezerra HG, Ozaki Y, Bruining N, Dudek D, Radu M, Erglis A, Motreff P, Alfonso F, Toutouzas K, Gonzalo N, Tamburino C, Adriaenssens T, Pinto F, Serruys PW, Di Mario C; Expert's OCT Review Document. Expert review document part 2: methodology, terminology and clinical applications of optical coherence tomography for the assessment of interventional procedures. Eur Heart J. 2012 Oct;33(20):2513-20. doi: 10.1093/eurheartj/ehs095. Epub 2012 May 31. No abstract available. PMID 22653335
- [Background] Tearney GJ, Regar E, Akasaka T, Adriaenssens T, Barlis P, Bezerra HG, Bouma B, Bruining N, Cho JM, Chowdhary S, Costa MA, de Silva R, Dijkstra J, Di Mario C, Dudek D, Falk E, Feldman MD, Fitzgerald P, Garcia-Garcia HM, Gonzalo N, Granada JF, Guagliumi G, Holm NR, Honda Y, Ikeno F, Kawasaki M, Kochman J, Koltowski L, Kubo T, Kume T, Kyono H, Lam CC, Lamouche G, Lee DP, Leon MB, Maehara A, Manfrini O, Mintz GS, Mizuno K, Morel MA, Nadkarni S, Okura H, Otake H, Pietrasik A, Prati F, Raber L, Radu MD, Rieber J, Riga M, Rollins A, Rosenberg M, Sirbu V, Serruys PW, Shimada K, Shinke T, Shite J, Siegel E, Sonoda S, Suter M, Takarada S, Tanaka A, Terashima M, Thim T, Uemura S, Ughi GJ, van Beusekom HM, van der Steen AF, van Es GA, van Soest G, Virmani R, Waxman S, Weissman NJ, Weisz G; International Working Group for Intravascular Optical Coherence Tomography (IWG-IVOCT). Consensus standards for acquisition, measurement, and reporting of intravascular optical coherence tomography studies: a report from the International Working Group for Intravascular Optical Coherence Tomography Standardization and Validation. J Am Coll Cardiol. 2012 Mar 20;59(12):1058-72. doi: 10.1016/j.jacc.2011.09.079. Erratum In: J Am Coll Cardiol. 2012 May 1;59(18):1662. Dudeck, Darius [corrected to Dudek, Darius]; Falk, Erlin [corrected to Falk, Erling]; Garcia, Hector [corrected to Garcia-Garcia, Hector M]; Sonada, Shinjo [corrected to Sonoda, Shinjo]; Troels, Thim [corrected to Thim, Troels]; van Es, Gerrit-Ann [correct. PMID 22421299
- [Background] Suzuki Y, Ikeno F, Koizumi T, Tio F, Yeung AC, Yock PG, Fitzgerald PJ, Fearon WF. In vivo comparison between optical coherence tomography and intravascular ultrasound for detecting small degrees of in-stent neointima after stent implantation. JACC Cardiovasc Interv. 2008 Apr;1(2):168-73. doi: 10.1016/j.jcin.2007.12.007. PMID 19463295
- [Background] Murata A, Wallace-Bradley D, Tellez A, Alviar C, Aboodi M, Sheehy A, Coleman L, Perkins L, Nakazawa G, Mintz G, Kaluza GL, Virmani R, Granada JF. Accuracy of optical coherence tomography in the evaluation of neointimal coverage after stent implantation. JACC Cardiovasc Imaging. 2010 Jan;3(1):76-84. doi: 10.1016/j.jcmg.2009.09.018. Epub 2010 Jan 12. PMID 20129535
- [Background] Templin C, Meyer M, Muller MF, Djonov V, Hlushchuk R, Dimova I, Flueckiger S, Kronen P, Sidler M, Klein K, Nicholls F, Ghadri JR, Weber K, Paunovic D, Corti R, Hoerstrup SP, Luscher TF, Landmesser U. Coronary optical frequency domain imaging (OFDI) for in vivo evaluation of stent healing: comparison with light and electron microscopy. Eur Heart J. 2010 Jul;31(14):1792-801. doi: 10.1093/eurheartj/ehq168. Epub 2010 Jun 5. PMID 20525979
- [Background] Gutierrez-Chico JL, van Geuns RJ, Regar E, van der Giessen WJ, Kelbaek H, Saunamaki K, Escaned J, Gonzalo N, di Mario C, Borgia F, Nuesch E, Garcia-Garcia HM, Silber S, Windecker S, Serruys PW. Tissue coverage of a hydrophilic polymer-coated zotarolimus-eluting stent vs. a fluoropolymer-coated everolimus-eluting stent at 13-month follow-up: an optical coherence tomography substudy from the RESOLUTE All Comers trial. Eur Heart J. 2011 Oct;32(19):2454-63. doi: 10.1093/eurheartj/ehr182. Epub 2011 Jun 9. PMID 21659439
- [Background] Toledano Delgado FJ, Alvarez-Ossorio MP, de Lezo Cruz-Conde JS, Bellido FM, Romero Moreno MA, Fernandez-Aceytuno AM, de Lezo Herrerosde Tejada JS, Pineda SO, Saint-Gerons JM, Pavlovic D. Optical coherence tomography evaluation of late strut coverage patterns between first-generation drug-eluting stents and everolimus-eluting stent. Catheter Cardiovasc Interv. 2014 Nov 1;84(5):720-6. doi: 10.1002/ccd.25235. Epub 2013 Oct 31. PMID 24174291
- [Background] Kim JS, Jang IK, Kim JS, Kim TH, Takano M, Kume T, Hur NW, Ko YG, Choi D, Hong MK, Jang Y. Optical coherence tomography evaluation of zotarolimus-eluting stents at 9-month follow-up: comparison with sirolimus-eluting stents. Heart. 2009 Dec;95(23):1907-12. doi: 10.1136/hrt.2009.167759. Epub 2009 Jun 16. PMID 19535352
- [Background] Chieffo A, Buchanan GL, Parodi G, Versaci F, Bianchi RM, Valenti R, Sacca S, Mongiardo A, Span S, Migliorini A, Spaccarotella C, Reimers B, Antoniucci D, Indolfi C, Ferrari A, Maehara A, Mintz GS, Colombo A. Drug-eluting stent implantation in patients with acute coronary syndrome - the Activity of Platelets after Inhibition and Cardiovascular Events: Optical Coherence Tomography (APICE OCT) study. EuroIntervention. 2014 Dec;10(8):916-23. doi: 10.4244/EIJY14M06_10. PMID 24974806
- [Background] Verheye S, Ormiston JA, Stewart J, Webster M, Sanidas E, Costa R, Costa JR Jr, Chamie D, Abizaid AS, Pinto I, Morrison L, Toyloy S, Bhat V, Yan J, Abizaid A. A next-generation bioresorbable coronary scaffold system: from bench to first clinical evaluation: 6- and 12-month clinical and multimodality imaging results. JACC Cardiovasc Interv. 2014 Jan;7(1):89-99. doi: 10.1016/j.jcin.2013.07.007. Epub 2013 Oct 16. PMID 24139932
- [Background] Kim JS, Jang IK, Fan C, Kim TH, Kim JS, Park SM, Choi EY, Lee SH, Ko YG, Choi D, Hong MK, Jang Y. Evaluation in 3 months duration of neointimal coverage after zotarolimus-eluting stent implantation by optical coherence tomography: the ENDEAVOR OCT trial. JACC Cardiovasc Interv. 2009 Dec;2(12):1240-7. doi: 10.1016/j.jcin.2009.10.006. PMID 20129551
- [Background] Qian J, Zhang YJ, Xu B, Yang YJ, Yan HB, Sun ZW, Zhao YL, Tang YD, Gao Z, Chen J, Cui JG, Mintz GS, Gao RL. Optical coherence tomography assessment of a PLGA-polymer with electro-grafting base layer versus a PLA-polymer sirolimus-eluting stent at three-month follow-up: the BuMA-OCT randomised trial. EuroIntervention. 2014 Nov;10(7):806-14. doi: 10.4244/EIJY14M07_17. PMID 25033105
- [Background] Prati F, Romagnoli E, Valgimigli M, Burzotta F, De Benedictis M, Ramondo A, Mehran R, Stella PR. Randomized comparison between 3-month Cre8 DES vs. 1-month Vision/Multilink8 BMS neointimal coverage assessed by OCT evaluation: the DEMONSTRATE study. Int J Cardiol. 2014 Oct 20;176(3):904-9. doi: 10.1016/j.ijcard.2014.08.031. Epub 2014 Aug 13. PMID 25171966
- [Background] Mauri L, Kereiakes DJ, Yeh RW, Driscoll-Shempp P, Cutlip DE, Steg PG, Normand SL, Braunwald E, Wiviott SD, Cohen DJ, Holmes DR Jr, Krucoff MW, Hermiller J, Dauerman HL, Simon DI, Kandzari DE, Garratt KN, Lee DP, Pow TK, Ver Lee P, Rinaldi MJ, Massaro JM; DAPT Study Investigators. Twelve or 30 months of dual antiplatelet therapy after drug-eluting stents. N Engl J Med. 2014 Dec 4;371(23):2155-66. doi: 10.1056/NEJMoa1409312. Epub 2014 Nov 16. PMID 25399658
- [Background] Colombo A, Chieffo A, Frasheri A, Garbo R, Masotti-Centol M, Salvatella N, Oteo Dominguez JF, Steffanon L, Tarantini G, Presbitero P, Menozzi A, Pucci E, Mauri J, Cesana BM, Giustino G, Sardella G. Second-generation drug-eluting stent implantation followed by 6- versus 12-month dual antiplatelet therapy: the SECURITY randomized clinical trial. J Am Coll Cardiol. 2014 Nov 18-25;64(20):2086-97. doi: 10.1016/j.jacc.2014.09.008. Epub 2014 Sep 15. PMID 25236346
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for Universal Definition of Myocardial Infarction; Authors/Task Force Members Chairpersons; Thygesen K, Alpert JS, White HD; Biomarker Subcommittee; Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA; ECG Subcommittee; Chaitman BR, Clemmensen PM, Johanson P, Hod H; Imaging Subcommittee; Underwood R, Bax JJ, Bonow JJ, Pinto F, Gibbons RJ; Classification Subcommittee; Fox KA, Atar D, Newby LK, Galvani M, Hamm CW; Intervention Subcommittee; Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J; Trials & Registries Subcommittee; Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML; Trials & Registries Subcommittee; Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G; Trials & Registries Subcommittee; Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D; Trials & Registries Subcommittee; Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG); Bax JJ, Baumgartner H, Ceconi C, Dean V, Deaton C, Fagard R, Funck-Brentano C, Hasdai D, Hoes A, Kirchhof P, Knuuti J, Kolh P, McDonagh T, Moulin C, Popescu BA, Reiner Z, Sechtem U, Sirnes PA, Tendera M, Torbicki A, Vahanian A, Windecker S; Document Reviewers; Morais J, Aguiar C, Almahmeed W, Arnar DO, Barili F, Bloch KD, Bolger AF, Botker HE, Bozkurt B, Bugiardini R, Cannon C, de Lemos J, Eberli FR, Escobar E, Hlatky M, James S, Kern KB, Moliterno DJ, Mueller C, Neskovic AN, Pieske BM, Schulman SP, Storey RF, Taubert KA, Vranckx P, Wagner DR. Third universal definition of myocardial infarction. J Am Coll Cardiol. 2012 Oct 16;60(16):1581-98. doi: 10.1016/j.jacc.2012.08.001. Epub 2012 Sep 5. No abstract available. PMID 22958960